CLINICAL TRIAL: NCT06220149
Title: FIT for Post poLypectomy bLeeding Prediction
Brief Title: Post Polypectomy Bleeding. Que Sera, Sera? Whatever Will be, Will be?
Acronym: FILLIP
Status: Recruiting | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Mihai Ciocirlan, Associate Professor of Gastroenterology, Carol Davila University of Medicine and Pharmacy
Other Study IDs: FILLIP
Record Dates: First submitted 2024-01-09; First posted 2024-01-23 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Polyp Colorectal; Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colorectal adenoma resected through different techniques (polypectomy, endoscopic mucosal resection, underwater endoscopic mucosal resection, endoscopic submucosal dissection)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post polypectomy cohort
  Interventions: Diagnostic Test: FIT (fecal immunochemical test)

INTERVENTIONS:
Diagnostic Test: FIT (fecal immunochemical test) — A FIT (fecal immunochemical test) will be done daily for the 14 days following polypectomy.

SUMMARY:
Patients with colorectal polyps removed endoscopically (polypectomy, endoscopic mucosal resection, underwater endoscopic mucosal resection, endoscopic submucosal dissection) may experience delayed post polypectomy bleeding. The incidence is about one in 40 cases.

There are risks factors for this complication, depending on the polyp type, patient demographics and co-morbidities and polypectomy technique. There are meta-analysis and nomograms for risk prediction available.

We will try to predict delayed post polypectomy bleeding by using FIT (fecal immunochemical test), with a cut-off adapted to detect post polypectomy bleeding, administered daily for 2 weeks after polypectomy.

DETAILED DESCRIPTION:
Why should one be concerned about delayed post polypectomy bleeding (DPPB)? One in 40 patients with polypectomy for large polyps will have it. A large systematic review of 50 studies including 6779 large polyps > 20mm resected by polypectomy, endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD), "en bloc" or in piece-meal have had an DPPB incidence of 2.6% (2.1% - 3.2%) [1].

Cand we generally predict what group of patients are more likely to have DPPB? Jaruvongvanich et al [2] have designed a meta-analysis of 12 studies on 14,313 patients. The pooled DPPB rate was 1.5% (0.7% - 3.4%). Cardiovascular disease (OR = 1.55), hypertension (OR = 1.53), polyp size > 10 mm (OR = 3.41), and polyps located in the right colon (OR = 1.60) were identified as significant DPPB risk factors, whereas age, sex, alcohol use, smoking, diabetes, cerebrovascular disease, pedunculated morphology, and carcinoma histology were not.

Huai et al [3] have designed a nomogram for DPPB prediction, based on 6 parameters, with a high AUC of 0.824 in the validation model, as in Figure 1, below. The model states that older men on anticoagulant, with pedunculated polyps on the right side are likely to bleed more often. Age, gender, and pedunculated morphology were included in the model, as risk factors, as opposed to previously mentioned paper [2]. The jury is probably still out for certain risk factors.

Yet, at the individual level, what could a patient do? Could a form of active surveillance for DPPB may be proposed?

Here's an idea. Fecal Immunochemical Test (FIT). FIT can detect minute quantities of hemoglobin in faces. It is used for colorectal cancer population screening in asymptomatic average risk individuals (eg. 50 to 75 years old) or in primary care in certain groups of symptomatic individuals, without overt rectal bleeding, as an adjunct decision tool for colonoscopy evaluation [5]. A recent meta-analysis on more than 6 million asymptomatic average risk individuals of which more than 2.6 million completed a screening FIT test have found a 5.4% positivity rate, an 85% colonoscopy completion rate, a 47.8% adenoma detection rate, a 25.3% advanced adenoma detection rate and a 5.1% colorectal cancer rate [6].

The fecal hemoglobin (f-Hb) cut-offs are set at 10 or 20 microg/g feces in majority of screening programs, depending on colorectal cancer incidence and the healthcare system's colonoscopy availability [7]. FIT result is usually read in central laboratory by specialized machines with cut-off threshold set by the health policy makers.

Mowat et al [8] have used FIT tests differently. They studied the dynamic of FIT values, before and after colonoscopy with polypectomy. They have found that the median pre-polypectomy f-Hb was significantly greater in advanced adenomas as compared to non-advanced adenomas (6.0 vs. 1.0 μg/g feces, p < 0.0001). For patients with both pre and post polypectomy FIT, the dynamic showed a significant decrease for advanced adenomas (19.2 microg/g pre-polypectomy decreasing to 3.5 microg/g post-polypectomy, p=0.01) and remained fairly constant and low for non-advanced adenomas (0.8 microg/g pre-polypectomy to 1.0 microg/g post-polypectomy, p = 0.96). To note that the authors recommended patients that the second FIT test be taken after 3-weeks to allow healing of colorectal resection site, an interval arbitrarily chosen based on experience. This would theoretically avoid false positive elevated quantitative FIT test values due to occult bleeding form the resection site.

Maybe we can use FIT for DPPB surveillance. There are, however, few obstacles:

* The time to epithelization of a resection site is unknown, possibly 3-weeks as Mowat et al [8] have assumed. It depends on lesion size and whether the resection site has been closed with metallic clips.
* The occult bleeding from the resection site depends on time to epithelization, the prophylactic coagulation of vessels at the end of the procedure (snare tip, APC, CoagGrasper), the use of hemostatic gel (Purastat).
* The probability of positive FIT depends on the occult bleeding from the resection site, location (rectum versus right colon) and FIT cut-off value.
* FIT laboratory central reading for quantitative tests takes a certain amount of time (post office time) which defies the purpose of a rapid result for an immediate individual predictive information.
* DPPB mostly occurs in the first week after polypectomy and extremely rarely in the second week after polypectomy [4].

There are a lot of known unknowns and unknown unknowns.

We propose to use a rapid qualitative FIT test to be self-administered daily by the patient in the first 2 weeks after colonoscopy, after each passage of feces.

This will hopefully identify a desirable dynamic pattern of FIT results:

* Positive daily until day X, negative afterwards
* Positive daily until day X, negative afterwards, but then again positive in day Y just before DPPB We could hypothetically, do a rapid test in the day Y and if negative maybe leave the patient go about his usual activities, hobbies, and holidays.

The proposed qualitative rapid FIT is HEMOTRUST (Biosyntex, Switzerland, www.biosyntex.com). The cut-off for HEMOTRUST is 6 microg/g, which is lower than advanced adenoma pre-polypectomy values and higher than post-polypectomy values for both advanced and non-advanced adenomas [8].

Aim of the research project We aim to study the DPPB predictive value of FIT after resection of advanced colorectal adenomas.

Question of the research project Is there a dynamic of f-Hb presence after resection of advanced adenomas? Is this dynamic different in patients with DPPB after resection of advanced adenomas? Could we predict DPPB by studying f-Hb dynamic using qualitative rapid FIT?

Hypothesis The f-Hb assessment dynamic using qualitative rapid FIT may help predict DPPB at the individual level.

ELIGIBILITY:
Inclusion Criteria:

* Patient with at least one advanced adenoma > 10mm diameter resected at colonoscopy by polypectomy, EMR, underwater EMR or ESD
* Age > 18 years old
* Written informed consent.

Exclusion Criteria:

* Synchronous advanced colorectal cancer
* Synchronous unresected advanced adenomas
* Concomitant inflammatory bowel disease or any active colitis
* Absence of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient above 18 years old with the indication of colonoscopy, satisfying inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Day of maximum probability of positive FIT to detect delayed post polypectomy bleeding | 14 days
  Day (1 - 14) of positive FIT with maximum 24h before delayed post polypectomy bleeding

SECONDARY OUTCOMES:
Time to delayed post polypectomy bleeding | 14 days
  Duration to delayed post polypectomy bleeding
Time of FIT positivity after polypectomy with no delayed post polypectomy bleeding | 14 days
  Duration of FIT positivity after polypectomy with no delayed post polypectomy bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- "Agrippa Ionescu" Hospital, Bucharest, Romania

REFERENCES:
- [Background] Hassan C, Repici A, Sharma P, Correale L, Zullo A, Bretthauer M, Senore C, Spada C, Bellisario C, Bhandari P, Rex DK. Efficacy and safety of endoscopic resection of large colorectal polyps: a systematic review and meta-analysis. Gut. 2016 May;65(5):806-20. doi: 10.1136/gutjnl-2014-308481. Epub 2015 Feb 13. PMID 25681402
- [Background] Jaruvongvanich V, Prasitlumkum N, Assavapongpaiboon B, Suchartlikitwong S, Sanguankeo A, Upala S. Risk factors for delayed colonic post-polypectomy bleeding: a systematic review and meta-analysis. Int J Colorectal Dis. 2017 Oct;32(10):1399-1406. doi: 10.1007/s00384-017-2870-0. Epub 2017 Aug 5. PMID 28779355
- [Background] Huai J, Ye X, Ding J. Nomogram for the Prediction of Delayed Colorectal Post-Polypectomy Bleeding. Turk J Gastroenterol. 2021 Sep;32(9):727-734. doi: 10.5152/tjg.2021.20842. PMID 34609301
- [Background] Lu Y, Zhou X, Chen H, Ding C, Si X. Establishment of a model for predicting delayed post-polypectomy bleeding: A real-world retrospective study. Front Med (Lausanne). 2022 Oct 19;9:1035646. doi: 10.3389/fmed.2022.1035646. eCollection 2022. PMID 36341244
- [Background] Monahan KJ, Davies MM, Abulafi M, Banerjea A, Nicholson BD, Arasaradnam R, Barker N, Benton S, Booth R, Burling D, Carten RV, D'Souza N, East JE, Kleijnen J, Machesney M, Pettman M, Pipe J, Saker L, Sharp L, Stephenson J, Steele RJ. Faecal immunochemical testing (FIT) in patients with signs or symptoms of suspected colorectal cancer (CRC): a joint guideline from the Association of Coloproctology of Great Britain and Ireland (ACPGBI) and the British Society of Gastroenterology (BSG). Gut. 2022 Jul 12;71(10):1939-62. doi: 10.1136/gutjnl-2022-327985. Online ahead of print. PMID 35820780
- [Background] Mohan BP, Khan SR, Daugherty E, Chandan S, Ponnada S, Facciorusso A, Kassab LL, Asokkumar R, Adler DG. Pooled rates of adenoma detection by colonoscopy in asymptomatic average-risk individuals with positive fecal immunochemical test: a systematic review and meta-analysis. Gastrointest Endosc. 2022 Aug;96(2):208-222.e14. doi: 10.1016/j.gie.2022.04.004. Epub 2022 Apr 9. PMID 35413330
- [Background] Pokharel R, Lin YS, McFerran E, O'Mahony JF. A Systematic Review of Cost-Effectiveness Analyses of Colorectal Cancer Screening in Europe: Have Studies Included Optimal Screening Intensities? Appl Health Econ Health Policy. 2023 Sep;21(5):701-717. doi: 10.1007/s40258-023-00819-3. Epub 2023 Jun 28. PMID 37380865
- [Background] Mowat C, Digby J, Cleary S, Gray L, Datt P, Goudie DR, Steele RJ, Strachan JA, Humphries A, Fraser CG. Faecal haemoglobin concentration in adenoma, before and after polypectomy, approaches the ideal tumour marker. Ann Clin Biochem. 2022 Jul;59(4):272-276. doi: 10.1177/00045632221080897. Epub 2022 Mar 2. PMID 35235491